CLINICAL TRIAL: NCT00839904
Title: The Effect of Physical Activity on the Mental and Physical Health of Children With Cancer in Remission
Brief Title: Physical Activity and Health of Children With Cancer in Remission
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Israel Cancer Association (Other)
Responsible Party: Principal Investigator, gal dubnov raz, Senior physician, Sheba Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GDR2-HMO-CTIL
Record Dates: First submitted 2009-02-08; First posted 2009-02-10 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Children; Cancer; Exercise
Keywords: children; cancer; exercise; fitness; body composition
MeSH Terms: conditions — Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- exercise (Experimental): two supervised, 60-minute weekly exercise sessions + instructions to perform additional physical activities throughout the day
  Interventions: Behavioral: exercise
- control (No Intervention): no intervention

INTERVENTIONS:
Behavioral: exercise — two supervised, 60-minute weekly exercise sessions + instructions to perform additional physical activities throughout the day
  Arms: exercise

SUMMARY:
Physical activity is a well-known and powerful tool in medicine,having preventive, palliative, and curative properties. This has not been sufficiently examined in children in remission from cancer. In this study, children in remission from cancer will be divided into exercise and control groups. The interventional group will perform two supervised, 60-minute weekly exercise sessions. Outcome measures of the exercise intervention will be quality of life, mood, cardiorespiratory fitness, body composition and bone mineral density.

ELIGIBILITY:
Inclusion Criteria:

* children aged 6-16
* remission from cancer
* >6 months after completion of all therapy

Exclusion Criteria:

* informed consent not given in writing
* refusal of tests: blood, fitness, questionnaires or DEXA
* locomotive handicaps
* extreme fatigue, nausea, dyspnea
* concurrent acute illness
* recent (less than 3 months) hospitalization
* documented (echocardiographic or nuclear medicine) decrease in cardiac function
* abnormal blood tests: Hb < 10 gr/dl, neutropenia < 500/mm3, thrombocytopenia < 50,000/mm3
* additional chronic health conditions unrelated to cancer (e.g. celiac disease, cerebral palsy, Down's syndrome)

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2010-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
health-related quality of life | 6months
mood | 6months
cardiorespiratory fitness | 6months
body fat percentage | 6months
bone mineral density | 6months